CLINICAL TRIAL: NCT04224727
Title: The Impact of Group Commitment Contracts on Smoking Cessation and Weight Loss
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was suspended due to low take-up in the group commitment contracts arm (~6%), revealing inadequate statistical power to justify moving forward. There were no safety concerns.
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0009
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation; Weight Loss
MeSH Terms: conditions — Smoking Cessation; Weight Loss

STUDY DESIGN:
Intervention Model Description: Respondents who meet the inclusion/exclusion criteria will be randomized into one of the following arms:
  1. Control Arm (No Intervention)
  2. Group Contract Arm
  3. Individual Monetary Rewards Arm
  4. Individual Commitment Contract Arm
  To understand the effect that knowledge about the effectiveness of commitment contracts has on uptake, smoking quit rates, and weight loss, we will be cross-randomizing those assigned to Arms #2-4 into further subgroups:
  Subgroup A. In the initial survey, participants will receive additional information treatments on the likelihood of success of the different incentives and contracts, with the goal of shifting "naives" to "sophisticates." In other words, we aim to provide information that will encourage present-biased or loss-averse individuals to participate in the programs that offer the greatest chance at success.
  Subgroup B. Participants will not receive any information about commitment contracts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control (No Intervention): Subjects are not offered a group commitment contract, individual commitment contract, or individual monetary rewards. Subjects do not receive additional information treatments.
- Group Commitment Contract + Information (Experimental): Subjects are offered a group commitment contract for smoking cessation or weight loss and receive additional information treatments.
  Interventions: Behavioral: Group Commitment Contract; Other: Information
- Individual Monetary Rewards + Information (Experimental): Subjects are offered individual monetary rewards for smoking cessation or weight loss and receive additional information treatments.
  Interventions: Behavioral: Individual Monetary Rewards; Other: Information
- Individual Commitment Contract + Information (Experimental): Subjects are offered an individual commitment contract for smoking cessation or weight loss and receive additional information treatments.
  Interventions: Behavioral: Individual Commitment Contract; Other: Information
- Group Commitment Contract (Experimental): Subjects are offered a group commitment contract for smoking cessation or weight loss and receive no additional information treatments.
  Interventions: Behavioral: Group Commitment Contract
- Individual Monetary Rewards (Experimental): Subjects are offered individual monetary rewards for smoking cessation or weight loss and receive no additional information treatments.
  Interventions: Behavioral: Individual Monetary Rewards
- Individual Commitment Contract (Experimental): Subjects are offered an individual commitment contract for smoking cessation or weight loss and receive no additional information treatments.
  Interventions: Behavioral: Individual Commitment Contract

INTERVENTIONS:
Behavioral: Group Commitment Contract — A group contract where the primary individual, who will be tracked by the study, can invite peers to join the contract and form their group. To initiate a contract, a user must choose: the stakes, start date, and (for weight loss contracts) target weight, and and, optionally, to allow other members to have the power to invite other people to join the group.
  Arms: Group Commitment Contract; Group Commitment Contract + Information
Behavioral: Individual Monetary Rewards — Individuals eligible for a $100 monetary reward (incentive) following verified smoking cessation or weight loss.
  Arms: Individual Monetary Rewards; Individual Monetary Rewards + Information
Behavioral: Individual Commitment Contract — Individuals will have the opportunity to create an individual commitment contract to quit smoking. They will have the option to set the stakes, start date, and (for weight loss contracts) target weight.
  Arms: Individual Commitment Contract; Individual Commitment Contract + Information
Other: Information — In the initial survey, participants will receive additional information treatments on the likelihood of success of the different incentives and contracts, with the goal of shifting "naives" to "sophisticates."
  Arms: Group Commitment Contract + Information; Individual Commitment Contract + Information; Individual Monetary Rewards + Information

SUMMARY:
We will conduct a randomized controlled trial to evaluate the effectiveness of group commitment contracts for smoking cessation and weight loss.

DETAILED DESCRIPTION:
Initial screening will be conducted online via the Qualtrics survey platform. Respondents meeting the inclusion/exclusion criteria will immediately be randomized into one of the intervention arms described below, and then take a baseline survey. This baseline survey will also be conducted online via the Qualtrics survey platform. The initial screening, randomization, and baseline survey should take approximately 15 minutes total and can be completed anywhere the participant has an internet connection.

INTERVENTION: Respondents who meet the inclusion/exclusion criteria will be randomized into one of the following arms:

1. Control Arm (No Intervention)
2. Group Contract Arm
3. Individual Monetary Rewards Arm
4. Individual Commitment Contract Arm

Subjects in Arms #2-4 will be cross-randomized into two subgroups:

A. Additional information treatments on the likelihood of success of the different incentives and contracts, with the goal of shifting "naives" to "sophisticates."

B. No additional information treatments.

FOLLOW-UP SURVEY: After the participants finish their contract, they will be emailed a link to the follow-up survey that will be administered online via the Qualtrics survey platform. The survey should take approximately 5 minutes and can be completed anywhere the participant has an internet connection. Participants will be directly prompted to answer whether they have been able to quit smoking or lose their target weight in the past six months. If a participant self-reports a claim of smoking cessation or successful weight loss, they will be asked to furnish at-home verification of their claim.

IN-PERSON VERIFICATION: A randomly selected subset of successful participants will be asked for in-person verification of their claim with a urine test (smoking cessation) or in-person weigh-in (weight loss) at a Quest Diagnostics location of their choice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Has smartphone with capability to reach internet daily and download app
* Able and willing to visit Quest location or take an at-home verification test
* Willing to furnish a payment method for commitment contract stakes

If completing a smoking cessation contract:

* Daily smoker

If completing a weight loss contract:

* Has access to a functioning scale
* Interest in losing weight at a pace of 2 lb or fewer per week, with a target BMI at or above 18.5

Exclusion Criteria:

* Pregnancy
* Any terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-06-19 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation / Weight Loss | 6 months
  Participants will be directly prompted to answer whether they have been able to quit smoking or reach their target weight in the past six months. If a participant self-reports a claim of success, they will be asked to furnish at-home (and, in some cases, in-person) verification.

OTHER OUTCOMES:
Smoking Cessation / Weight Loss by Sex/Gender, Race, and Ethnicity | 6 months
  Participants will be directly prompted to answer whether they have been able to quit smoking or reach their target weight in the past six months. If a participant self-reports a claim of success, they will be asked to furnish at-home (and, in some cases, in-person) verification.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Karlan, PhD, Principal Investigator — Northwestern University; Anna Tuchman, PhD, Principal Investigator — Northwestern University; Jonathan Zinman, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Northwestern University, Global Poverty Research Lab, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code